CLINICAL TRIAL: NCT01300858
Title: A Phase I/II Study of the Safety and Biological Activity of Intraperitoneal EGEN-001 (IL-12 Plasmid Formulated With PEG-PEI-Cholesterol Lipopolymer) Administered Alone and in Combination With Standard Chemotherapy in Colorectal Peritoneal Carcinomatosis Patients Who Had Previously Received Cytoreductive Surgery Plus Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Therapy
Brief Title: A Study of the Safety and Biological Activity of Intraperitoneal (IP) EGEN-001 Administered Alone and in Combination With Standard Chemotherapy in Colorectal Peritoneal Carcinomatosis Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sites could not enroll patients.
Sponsor: EGEN, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGEN-001-301
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EGEN-001 (Experimental)
  Interventions: Drug: EGEN-001-301

INTERVENTIONS:
Drug: EGEN-001-301 — Patients will be treated with EGEN-001 intra-peritoneally (IP) once every week for 12 weeks and then once every two weeks until disease progression or intolerable toxicity, but for no more than one year. Patients who develop progressive metastases will receive standard chemotherapy concomitant with EGEN-001. Hence, the initial EGEN-001 treatment period will be without chemotherapy. The standard chemotherapy regimen will be FOLFOX or FOLFIRI administered every 2-3 weeks. Patient with progressive disease a second time will be taken off-study. Those who remain progression-free will receive EGEN-001 for up to one year.

SUMMARY:
Colorectal cancer may be caused by a build-up of genetic defects, or damaged genes within the body's cells. When genes are damaged, the body may be unable to produce a group of proteins, called cytokines, used by the immune system to fight cancer and some infections. The investigational gene transfer agent EGEN-001 contains the human gene for the cytokine interleukin-12 (IL-12) in a special carrier system designed to enter the cells and help the body to produce cytokines.Therefore Therefore, the purpose of the EGEN-001 therapy is to attempt to enhance the body's natural ability to recognize and fight cancer cells.

DETAILED DESCRIPTION:
This multi-center, Phase I/II study will be conducted with an open-label, non-randomized design. The study will enroll up to 30 patients who had gone through cytoreductive surgery and HIPEC treatment 6-8 weeks prior to enrollment. Patients will be treated with EGEN-001 24 mg/m2 intra-peritoneally (IP) once every week for 12 weeks and then once every two weeks until disease progression or intolerable toxicity, but for no more than one year. Patients who develop progressive metastases will receive standard chemotherapy concomitant with EGEN-001. Hence, the initial EGEN-001 treatment period will be without chemotherapy. The standard chemotherapy regimen will be FOLFOX or FOLFIRI administered every 2-3 weeks. Patient with progressive disease a second time will be taken off-study. Those who remain progression-free will receive EGEN-001 for up to one year.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age (or minimum legal age and competency to provide voluntary written informed consent for study participation) and no more than 80 years of age.
* Patients must have colorectal carcinoma (including appendiceal) with metastases limited to peritoneal cavity. Histological documentation of the original primary tumor is required via pathology report.
* Patients must have completed surgical debulking + hyperthermic intraperitoneal chemotherapy (mitomycin) and have had a peritoneal catheter inserted 6-8 weeks before beginning infusion with IP EGEN-001 and must have post-debulking peritoneal cancer index (PCI) of <2. Patients do not have to have measurable metastases by RECIST criteria following surgical debulking.
* Patients may have received previous systemic chemotherapy for colorectal cancer, but this is not required.
* Patients must have an ECOG Performance Status of 0, 1, or 2.
* Any other prior therapy directed at the malignant tumor, including biological and immunologic agents, must be discontinued at least three weeks prior to enrollment.
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated UTI.)
* Patients must have adequate:

  1. Bone marrow function: Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl, equivalent to the Active Version of the NCI Common Terminology Criteria (CTCAE) grade 1. Platelets greater than or equal to 100,000/mcl.
  2. Renal function: creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), per the Active Version of the NCI CTCAE grade 1.
  3. Hepatic function: Bilirubin less than or equal to 1.5 x ULN (per the Active Version of the NCI CTCAE grade 1). SGOT (AST) less than or equal to 3 x ULN (per the Active Version of the NCI CTCAE grade 1) and alkaline phosphatase less than or equal to 2.5 x ULN (per the Active Version of the NCI CTCAE grade 1).
  4. Neurologic function: Neuropathy (sensory and motor) less than or equal to the Active Version of the NCI CTCAE grade 1.
* Patients must have signed an approved informed consent and authorization permitting release of personal health information.
* Women of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception. Female partners of childbearing potential of male patients must also use an effective form of contraception. Contraception must be used for 90 days following the last dose of EGEN-001.

Exclusion Criteria:

* Patients who have had prior therapy with EGEN-001 or IL-12.
* Prior radiation therapy to the abdomen or pelvis less than 6 months prior to entering the study.
* Patients with a serious uncontrolled medical illness or disorder or active infection within four weeks of study entry.
* Patients with any condition/anomaly that would interfere with the appropriate placement of the IP catheter for study drug administration including: intestinal dysfunction or suspected extensive adhesions from prior history or finding at laparoscopy.
* Metastases beyond the peritoneal cavity including liver, lung or retroperitoneal lymph nodes.
* History of other malignancy other than non-melanoma skin cancer or in situ cervical carcinoma within the last 5 years.
* The patient is pregnant or lactating.
* The patient has taken an investigational agent in the preceding 4 weeks.
* Patients with a history of HIV, hepatitis B or hepatitis C.
* Patients who require treatment with pharmacologic doses of systemic steroids; replacement doses, topical, inhalation and ophthalmic steroid use is permitted.
* Patients who are allergic to any of the components of EGEN-001.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 5 years
Overall survival | 5 years
Tumor Growth Assessment by X-ray/CT | 1 year

SECONDARY OUTCOMES:
Number of study subjects with adverse events | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Midwestern Regional Medical Center, Zion, Illinois, United States